CLINICAL TRIAL: NCT01197937
Title: Relationship of Realize Mysuccess Usage to Outcomes of Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Ethicon Endo-Surgery (Industry)
Responsible Party: Principal Investigator, David Sarwer, Professor of Psychology in Psychiatry and Surgery at The Perelman School of Medicine, University of Pennsylvania
Other Study IDs: 29372
Record Dates: First submitted 2010-09-02; First posted 2010-09-09 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Bariatric Surgery; Obesity; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this observational study is to assess the efficacy of Realize My Success (RMS),a website that allows patients and providers to maintain contact via the website. We will compare RMS users on a number of different variables with the goal of identifying which variables are associated with optimal outcomes (larger weight losses) at one year (and potentially beyond). The study has two primary objectives. The first is to assess changes in body weight at postoperative year 1 in frequent v. infrequent RMS users. We predict that frequent users will achieve significantly greater reductions in weight at 6 and 12 months (and beyond) than infrequent users. The second objective is to assess changes in body weight at postoperative year 1 in persons who use different features of the RMS site. We hypothesize that persons who, on a regular basis, record their food intake, track their physical activity and make specific behavioral goals will experience significantly greater reductions in weight beginning 6 months after surgery as compared to those who do not use these features of the RMS site.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* BMI between 40-70 kg/m2 (or 35-70 kg/m2 in the presence of co-morbidities)
* Have registered in the Realize Mysuccess Systema and have logged into the system at least once postoperatively.

Exclusion Criteria:

* We will be receiving/analyzing a data set based on the inclusion criteria, therefore there is no set exclusion criteria for our research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be men and women, 18-65 years old, with a BMI of 40-70 kg/m2 (or 35-70 kg/m2 in the presence of co-morbidities) who have registered in the RMS system and have log into the system at least once postoperatively.
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Actual)
Dates: Start 2010-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Assess changes in body weight in frequent v. infrequent RMS users | 12 months